CLINICAL TRIAL: NCT03230643
Title: Evaluation of Baroreflex Activation Therapy in Patients With Advanced Heart Failure
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: HDZ-KA_012_DG
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Barostim neo implantation — The Barostim neo Implantation is a new promising treatment option for patients with advanced heart failure (HEFrEF) as it might improve cardiac and vascular function by restoring sympathovagal-balance through its effects on the autonomic nervous system.
  In this observational study, data from patients who have received the Barostim neo System as part of clinical routine will be collected and analyzed. The implantation of this new device is not part of the study.

SUMMARY:
The objective of this single center prospective clinical trial is to evaluate the safety and efficacy of carotid Baroreflex Activation Therapy (BAT) in advanced heart failure (HFrEF). Beyond that, the primary aim of this study is to identify patients of the whole HFrEF population that are most likely to benefit from this new promising therapy.

DETAILED DESCRIPTION:
Baroreflex activation therapy (BAT) is a new treatment option for patients (pts) suffering from heart failure with reduced left ventricular ejection fraction (HFrEF) to improve functional status and quality of life. Yet it is unknown which pts of the whole HFrEF population are most likely to benefit from this new promising therapy. As this invasive technique should definitely not be proposed for all HFrEF pts with left ventricular ejection fraction of 35 % or less the aim of this single center prospective clinical trial is to evaluate to which extent possible factors (e.g. cardiac resynchronization therapy (CRT), atrial fibrillation) may influence the response to BAT. To analyze any possible differences concerning the modulation of the autonomic nervous system caused by BAT in the presence of atrial fibrillation or cardiac resynchronization therapy, heart rate variability (HRV) analyses will be performed additionally. As autonomic nervous activity plays a pivotal role in the genesis and termination of atrial fibrillation any possible impact of baroreflex activation therapy on atrial fibrillation will be examined.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure (NYHA functional class III)
* LVEF of 35% or less
* chronic stable Guideline-directed medical therapy (diuretic agent, angiotensin-converting enzyme inhibitor or angiotensin receptor blocker and a beta blocker, if tolerated)
* resting heart rate between 60 and 100 beats/min
* systolic blood pressure of at least 100 mmHg

Exclusion Criteria:

* estimated glomerular filtration rate < 30 ml/min/1.73 m²
* Plaque and atherosclerosis reducing the linear diameter of the internal or distal common carotid arteries by 50% or more
* acute pulmonary edema within the last six weeks
* implantation of Pacemakers, ICDs or CRTs within the last 3 months or planned for the next three months
* life expectancy < 1 year
* body mass index > 40 kg/m²
* symptomatic uncontrolled bradyarrhythmias
* severe asthma, chronic obstructive pulmonary disease or restrictive lung disease
* active malignancy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffering from advanced heart failure with left ventricular ejection fraction of 35 % or less are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction | measured baseline and during follow up visits 3, 6 and 12 months after inclusion or Baroreflex Activation Therapy device activation
Change in Quality of life | assessed baseline and during follow up visits 3, 6 and 12 months after inclusion or Baroreflex Activation Therapy device activation
Change in NYHA functional class ranking | measured baseline and during follow up visits 3, 6 and 12 months after inclusion or Baroreflex Activation Therapy device activation
Chance in exercise capacity (distance walked in 6 min) | measured baseline and during follow up visits 3, 6 and 12 months after inclusion or Baroreflex Activation Therapy device activation
Change in N-terminal pro-brain natriuretic peptide | measured baseline and during follow up visits 3, 6 and 12 months after inclusion or Baroreflex Activation Therapy device activation

CONTACTS AND LOCATIONS:
Locations (1):
- Herz- und Diabeteszentrum NRW, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] DeMazumder D, Kass DA, O'Rourke B, Tomaselli GF. Cardiac resynchronization therapy restores sympathovagal balance in the failing heart by differential remodeling of cholinergic signaling. Circ Res. 2015 May 8;116(10):1691-9. doi: 10.1161/CIRCRESAHA.116.305268. Epub 2015 Mar 2. PMID 25733594
- [Result] Gronda E, Seravalle G, Trevano FQ, Costantino G, Casini A, Alsheraei A, Lovett EG, Vanoli E, Mancia G, Grassi G. Long-term chronic baroreflex activation: persistent efficacy in patients with heart failure and reduced ejection fraction. J Hypertens. 2015 Aug;33(8):1704-8. doi: 10.1097/HJH.0000000000000603. PMID 26132760
- [Result] Abraham WT, Zile MR, Weaver FA, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Little WC. Baroreflex Activation Therapy for the Treatment of Heart Failure With a Reduced Ejection Fraction. JACC Heart Fail. 2015 Jun;3(6):487-496. doi: 10.1016/j.jchf.2015.02.006. Epub 2015 May 14. PMID 25982108
- [Result] Zile MR, Abraham WT, Weaver FA, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Little WC. Baroreflex activation therapy for the treatment of heart failure with a reduced ejection fraction: safety and efficacy in patients with and without cardiac resynchronization therapy. Eur J Heart Fail. 2015 Oct;17(10):1066-74. doi: 10.1002/ejhf.299. Epub 2015 Jun 10. PMID 26011593
- [Result] Fantoni C, Raffa S, Regoli F, Giraldi F, La Rovere MT, Prentice J, Pastori F, Fratini S, Salerno-Uriarte JA, Klein HU, Auricchio A. Cardiac resynchronization therapy improves heart rate profile and heart rate variability of patients with moderate to severe heart failure. J Am Coll Cardiol. 2005 Nov 15;46(10):1875-82. doi: 10.1016/j.jacc.2005.06.081. Epub 2005 Oct 24. PMID 16286175
- [Result] Oliveira M. Comment on "Baroreflex Activation Therapy for the Treatment of Heart Failure With a Reduced Ejection Fraction". Rev Port Cardiol. 2015 Dec;34(12):795-7. doi: 10.1016/j.repce.2015.12.014. PMID 27099884
- [Result] Huang JH, Lin YK, Hsieh MH, Chen SA, Chiu WC, Chen YJ. Modulation of Autonomic Nervous Activity in the Termination of Paroxysmal Atrial Fibrillation. Pacing Clin Electrophysiol. 2017 Apr;40(4):401-408. doi: 10.1111/pace.13045. Epub 2017 Mar 3. PMID 28181276
- [Result] Linz D, Hohl M, Khoshkish S, Mahfoud F, Ukena C, Neuberger HR, Wirth K, Bohm M. Low-Level But Not High-Level Baroreceptor Stimulation Inhibits Atrial Fibrillation in a Pig Model of Sleep Apnea. J Cardiovasc Electrophysiol. 2016 Sep;27(9):1086-92. doi: 10.1111/jce.13020. Epub 2016 Jun 22. PMID 27235276
- [Result] Linz D, Mahfoud F, Schotten U, Ukena C, Neuberger HR, Wirth K, Bohm M. Effects of electrical stimulation of carotid baroreflex and renal denervation on atrial electrophysiology. J Cardiovasc Electrophysiol. 2013 Sep;24(9):1028-33. doi: 10.1111/jce.12171. Epub 2013 May 2. PMID 23638844
- [Result] Dai M, Bao M, Zhang Y, Yu L, Cao Q, Tang Y, Huang H, Wang X, Hu D, Huang C. Low-level carotid baroreflex stimulation suppresses atrial fibrillation by inhibiting left stellate ganglion activity in an acute canine model. Heart Rhythm. 2016 Nov;13(11):2203-2212. doi: 10.1016/j.hrthm.2016.08.021. Epub 2016 Aug 9. PMID 27520541